CLINICAL TRIAL: NCT07242417
Title: A Preliminary Clinical Study of TC-G203 for Patients With GPC3-Positive Recurrent/Metastatic Solid Tumors
Brief Title: TC-G203 for Patients With GPC3-Positive Advanced Solid Tumors
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Beijing GoBroad Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G203-IIT-01
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Solid Cancer; GPC3 Positive Hepatocellular Carcinoma
Keywords: Solid Cancer; GPC3 positive hepatocellular carcinoma
MeSH Terms: interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TC-G203 Cell Therapy (Experimental): TC-G203 CAR-T Cells Following lymphodepletion chemotherapy, participants will receive TC-G203 CAR-T cell infusion.
  Interventions: Biological: TC-G203 cells treatment

INTERVENTIONS:
Biological: TC-G203 cells treatment — TC-G203 CAR-T cells Treatment follows a lymphodepletion Drug: Fludarabine and Cyclophosphamide.
  Other Names: Cyclophosphamide; Fludarabine

SUMMARY:
This is a single-arm, open-label, dose-escalation clinical trial designed to evaluate the safety, tolerability, expansion, and persistence of TC-G203 in patients with GPC3-positive recurrent or metastatic solid tumors who have progressed after prior therapies. The primary objective is to determine the maximum tolerated dose (MTD), with a secondary aim to assess preliminary clinical efficacy in solid tumors.

DETAILED DESCRIPTION:
This study is designed as a single-arm, open-label, single-dose clinical trial to evaluate the safety and efficacy of TC-G203 therapy in patients with recurrent or metastatic solid tumors. The study protocol consists of five main stages: (1) patient screening, (2) collection of peripheral blood mononuclear cells (PBMCs), (3) lymphodepletion chemotherapy, (4) TC-G203 infusion, and (5) post-infusion follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must voluntarily provide written informed consent.
2. Aged 18-75 years (inclusive).
3. Life expectancy ≥ 12 weeks.
4. ECOG performance status 0-1.
5. Failed or unsuitable for standard therapy.
6. At least one measurable lesion per RECIST 1.1.
7. GPC3-positive tumor confirmed by immunohistochemistry.
8. Adequate organ and bone marrow function.
9. Effective contraception required for participants of childbearing potential.
10. Adequate venous access for leukapheresis.

Exclusion Criteria:

1. Primary CNS malignancy or uncontrolled CNS metastases.
2. Other malignancies within 5 years
3. Active autoimmune disease or history of autoimmune disease.
4. Immunodeficiency, including HIV positivity
5. Bleeding disorders (inherited or acquired).
6. Clinically significant cardiovascular disease.
7. Active infection (including tuberculosis, hepatitis C, syphilis).
8. Pregnant or breastfeeding women.
9. Severe systemic or psychiatric illness.
10. Prior cell or gene therapy.
11. Severe drug hypersensitivity history.
12. Investigator-assessed unsuitability for trial participation. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLT) and Maximum Tolerated Dose (MTD) | Within 28 days after TC-G203 infusion
  DLT is defined as any CAR-T cell-related adverse event graded per ASTCT 2019 CRS criteria and NCI CTCAE v5.0, including: ≥Grade 4 hematologic toxicity not recovering to ≤Grade 2 by Day 28, ≥Grade 4 CRS lasting ≥3 days, ≥Grade 3 ICANS, or ≥Grade 3 non-hematologic toxicity lasting >7 days (excluding fever, fatigue, nausea/vomiting).

SECONDARY OUTCOMES:
Tumor Response and Survival Outcomes | Up to 24 months
  Objective Response Rate (ORR): Number of participants with complete response (CR) or partial response (PR) Duration of Response (DOR): Time from first documented response to disease progression or death Progression-Free Survival (PFS): Time from TC-G203 infusion to disease progression or death Overall Survival (OS): Time from TC-G203 infusion to death from any cause

OTHER OUTCOMES:
Duration of Persistence of TC-G203 in Peripheral Blood | Up to 24 months
  Persistence of TC-G203 CAR-T cells in peripheral blood over time measured by qPCR and flow cytometry
Concentration of Pro-inflammatory Cytokines and Tumor Markers in Peripheral Blood | Up to 24 months
  Serum levels of IL-6, TNF-α, IL-8, IFN-γ, CRP, AFP, and sGPC3 at specified time points

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Gobroad Hospital, Beijing, Beijing Municipality
  - GoBroad Healthcare Group, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No